CLINICAL TRIAL: NCT01469832
Title: A Phase I/II, Open-Label, Multi-Center, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (hESC-RPE) Cells in Patients With Stargardt's Macular Dystrophy (SMD)
Brief Title: Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (hESC-RPE) Cells in Patients With Stargardt's Macular Dystrophy (SMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Institute for Regenerative Medicine (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7316-CL-0003; 2011-000054-34 (EudraCT Number); ACT hESC-RPE SMD 01 EU (Other: Sponsor)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Stargardt's Macular Dystrophy
Keywords: fundus flavimaculatus; Retinal Diseases; Macular Degeneration; SMD; juvenile macular dystrophy
MeSH Terms: conditions — Stargardt Disease; Retinal Diseases; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subretinal injection of MA09-hRPE (Experimental): * Cohort 1 50,000 cells
  * Cohort 2 100,000 cells
  * Cohort 2a Better Vision 100,000 cells
  * Cohort 3 150,000 cells
  * Cohort 4 200,000 cells
  Interventions: Biological: MA09-hRPE

INTERVENTIONS:
Biological: MA09-hRPE — * Cohort 1 50,000 cells
  * Cohort 2 100,000 cells
  * Cohort 2a Better Vision 100,000 cells
  * Cohort 3 150,000 cells
  * Cohort 4 200,000 cells

SUMMARY:
The purpose of this study is:

To evaluate the safety and tolerability of RPE cellular therapy in patients with SMD .

To evaluate potential efficacy endpoints to be used in future studies RPE cellular therapy.

DETAILED DESCRIPTION:
This study is a Phase I/II, open-label, non randomized, sequential, multi-center clinical trial. There will be 5 cohorts, the 4 low vision cohorts will contain 3 patients, the better vision cohort will contain 4 patients. The enrolled cohorts will be as follows:

Three SMD patients- 50,000 MA09-hRPE cells transplanted

Three SMD patients- 100,000 MA09-hRPE cells transplanted

Four Better Vision SMD patients- 100,000 MA09-hRPE cells transplanted

Three SMD patients- 150,000 MA09-hRPE cells transplanted

Three SMD patients- 200,000 MA09-hRPE cells transplanted

Patients will be enrolled sequentially, and within each cohort of 3 patients, each patient's clinical course over the first 6 weeks following cell transplantation will be reviewed by an independent (DSMB) before enrollment is opened for the next 2 patients. A full safety assessment of all 3 patients in each cohort will be made by the DSMB when the 3rd patient in each cohort completes 4 weeks of follow-up, and before the first patient in the next cohort receives a cell transplant. The exception is the better vision group where all patients may be enrolled once DSMB approval has been received.

Each cohort will be enrolled sequentially in turn, with the exception of the better vision cohort which may be enrolled in parallel with the other cohorts.

The day of the cell implantation will be Day 0, and patients will remain in the study until the last visit at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over 18 years of age. Clinical diagnosis of SMD If known, the patient"s genotype will be recorded in the medical history, if unknown, patient will allow for the submission of a sample for genotyping.

Independently verified clinical findings consistent with SMD. The visual acuity of the eye to receive the transplant will be no better than 20/400. The visual acuity of the eye in the better vision cohort to receive the transplant will be no better than 20/100.

The visual acuity of the eye that is not to receive the transplant will be no better than 20/400 for the worse vision patients and no worse than 20/100 for the better vision patients.

Electrophysiological findings consistent with SMD . Medically suitable to undergo vitrectomy and subretinal injection. Medically suitable for general anaesthesia or waking sedation, if needed.

Medically suitable for transplantation of an embryonic stem cell line:

* Normal serum chemistry (sequential multi-channel analyzer 20 [SMA-20]) and hematology (complete blood count [CBC], prothrombin time [PT], and activated partial thromboplastin time [aPTT]) screening tests.
* Negative urine screen for drugs of abuse.
* Negative human immunodeficiency virus (HIV), hepatitis B (HBV), and hepatitis C (HCV) serologies.
* No history of malignancy, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin.
* Negative cancer screening within previous 6 months:

complete history & physical examination; dermatological screening exam for malignant lesions; negative fecal occult blood test negative chest roentgenogram (CXR); normal CBC & manual differential; negative urinalysis (U/A);normal thyroid exam and thyroid panel; if male, normal testicular examination; if over age 40, digital rectal examination (DRE) and prostate specific antigen (PSA); if female, normal pelvic examination with Papanicolaou smear; and if female, normal clinical breast exam and if 50 years of age or older, negative mammogram.

If female and of childbearing potential, willing to use an effective form of birth control during the study.

If male, willing to use barrier and spermicide contraception during the study. Willing to defer all future blood, blood component or tissue donation. Able to understand and willing to sign the informed consent.

Exclusion Criteria:

* History of malignancy, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin.

History of myocardial infarction in previous 12 months. History of diabetes mellitus. Any immunodeficiency. Any current immunosuppressive therapy other than intermittent or low dose corticosteroids.

Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV. Current participation in any other clinical trial. Participation within previous 6 months in any clinical trial of a drug by ocular or systemic administration.

Any other sight-threatening ocular disease. Any chronic ocular medications. Any history of retinal vascular disease (compromised blood-retinal barrier. Glaucoma. Uveitis or other intraocular inflammatory disease. Significant lens opacities or other media opacity. Ocular lens removal within previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12-13 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
safety and tolerance of transplantation | 12 months
  The safety and tolerance of transplantation of hESC-derived MA09-hRPE will be considered safe and tolerated in the absence of: Any grade 2 NCI grading system)or greater adverse event related to the cell product.Any evidence that the cells are contaminated with an infectious agent, or have tumorigenic potential, Adverse Event and Serious Adverse Event assessment, Serial vital signs and Clinical laboratory tests Direct ophthalmological monitoring Monitoring of RPE cells acceptance/integrity/rejection Monitoring of local and systemic infection or tumorigenic cell transformation

SECONDARY OUTCOMES:
Evidence of successful engraftment | 12 months
  •Evidence of successful engraftmentEvidence of successful engraftment will consist of:
  * Structural evidence (OCT imaging, fluorescein angiography, autofluorescence photography, slit-lamp examination with fundus photography) that cells have been implanted in the correct location
  * Electroretinographic evidence (mfERG) showing enhanced activity in the implant location

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Institute for Regenerative Medicine
Locations (3):
- United Kingdom (3):
  - Lothian Health Board Headquarters at Waverley Gate, Edinburgh
  - Moorefields Eye Hospital NHS Foundation Trust, London
  - Newcastle on Tyne NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Background] Schwartz SD, Hubschman JP, Heilwell G, Franco-Cardenas V, Pan CK, Ostrick RM, Mickunas E, Gay R, Klimanskaya I, Lanza R. Embryonic stem cell trials for macular degeneration: a preliminary report. Lancet. 2012 Feb 25;379(9817):713-20. doi: 10.1016/S0140-6736(12)60028-2. Epub 2012 Jan 24. PMID 22281388
- [Background] Schwartz SD, Regillo CD, Lam BL, Eliott D, Rosenfeld PJ, Gregori NZ, Hubschman JP, Davis JL, Heilwell G, Spirn M, Maguire J, Gay R, Bateman J, Ostrick RM, Morris D, Vincent M, Anglade E, Del Priore LV, Lanza R. Human embryonic stem cell-derived retinal pigment epithelium in patients with age-related macular degeneration and Stargardt's macular dystrophy: follow-up of two open-label phase 1/2 studies. Lancet. 2015 Feb 7;385(9967):509-16. doi: 10.1016/S0140-6736(14)61376-3. Epub 2014 Oct 15. PMID 25458728
- [Derived] Mehat MS, Sundaram V, Ripamonti C, Robson AG, Smith AJ, Borooah S, Robinson M, Rosenthal AN, Innes W, Weleber RG, Lee RWJ, Crossland M, Rubin GS, Dhillon B, Steel DHW, Anglade E, Lanza RP, Ali RR, Michaelides M, Bainbridge JWB. Transplantation of Human Embryonic Stem Cell-Derived Retinal Pigment Epithelial Cells in Macular Degeneration. Ophthalmology. 2018 Nov;125(11):1765-1775. doi: 10.1016/j.ophtha.2018.04.037. Epub 2018 Jun 5. PMID 29884405
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;7316-CL-0003
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217491&parentIdentifier=7316-CL-0003&attachmentIdentifier=f0a212f7-4d32-484f-a92f-26ff8c4d318a&fileName=7316-CL-0003_0006_Plain_language_summary.pdf&versionIdentifier=